CLINICAL TRIAL: NCT04096638
Title: A Phase 1a/1b Dose-escalation Study of Intravenously Administered SB 11285 Alone and in Combination With Atezolizumab in Patients With Advanced Solid Tumors
Brief Title: Safety and Efficacy of SB 11285 Alone and in Combination With Atezolizumab in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: invoX Pharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBP-11285-ONC-101
Record Dates: First submitted 2019-09-03; First posted 2019-09-20 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-03

CONDITIONS: Melanoma; Head and Neck Squamous Cell Carcinoma; Solid Tumor
MeSH Terms: conditions — Melanoma; Squamous Cell Carcinoma of Head and Neck | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1a: Monotherapy Dose Escalation (Experimental): SB 11285 weekly on Days 1, 8, 15 and 22 on repeated 28-day cycles in escalating doses
  Interventions: Drug: SB 11285
- Part 1b: PD-L1 Combination Dose Escalation (Experimental): SB 11285 weekly on Days 1, 8, 15 and 22 on repeated 28-day cycles in escalating doses plus 1680mg every 4 weeks (Q4W) atezolizumab
  Interventions: Drug: SB 11285; Drug: Atezolizumab
- Part 2: Combination Expansion Cohorts at RP2D (Cohort A) (Experimental): Cohort A: Patients with Melanoma
  After determination of maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) in SB 11285 plus atezolizumab combination the Part 2 with expansion cohorts will commence to further evaluate the RP2D.
  Interventions: Drug: SB 11285; Drug: Atezolizumab
- Part 2: Combination Expansion Cohorts at RP2D (Cohort B) (Experimental): Cohort B: Patients with HNSCC
  After determination of maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) in SB 11285 plus atezolizumab combination the Part 2 with expansion cohorts will commence to further evaluate the RP2D.
  Interventions: Drug: SB 11285; Drug: Atezolizumab
- Part 2: Combination Expansion Cohorts at RP2D (Cohort C) (Experimental): Cohort C: Patients with tumor types other then Cohort A and B (Naïve or relapsed refractory to anti PD-1/PD-L1)
  After determination of maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) in SB 11285 plus atezolizumab combination the Part 2 with expansion cohorts will commence to further evaluate the RP2D.
  Interventions: Drug: SB 11285; Drug: Atezolizumab

INTERVENTIONS:
Drug: SB 11285 — SB 11285 2mg lyophilized powder for IV infusion
Drug: Atezolizumab — 1680 mg every 4 weeks
  Other Names: Tecentriq
  Arms: Part 1b: PD-L1 Combination Dose Escalation; Part 2: Combination Expansion Cohorts at RP2D (Cohort A); Part 2: Combination Expansion Cohorts at RP2D (Cohort B); Part 2: Combination Expansion Cohorts at RP2D (Cohort C)

SUMMARY:
A Phase 1a/1b, multicenter, open-label, non-randomized, dose-escalation, and cohort expansion study to examine the DLTs, MTD, and RP2D of SB 11285 administered as an IV infusion in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Part 1a of the study will assess the safety and tolerability of SB 11285 as monotherapy in eligible patients with advanced solid tumors. Part 1b will assess the safety and tolerability of SB 11285 in combination with atezolizumab in patients with advanced solid tumors. RP2D decisions will be based on the totality of data, including DLTs, tolerability, PK, pharmacodynamics, and efficacy, as available. Part 2 will further evaluate the combination RP2D of SB 11285 and atezolizumab in selected tumor types. Both Parts 1a and 1b of the study will use a standard 3+3 dose-escalation design with the dose escalated in successive cohorts of 3 to 6 patients each within each cohort in an open-label fashion. In Part 1a Monotherapy Dose Escalation, patients who meet eligibility criteria will receive IV SB 11285 as monotherapy weekly on Days 1, 8, 15, and 22 of repeated 28-day cycles in escalating doses. Once Dose Level 2 of Part 1a monotherapy have been evaluated by the Safety Review Committee (SRC) and have been declared to be safe to dose escalate to Dose Level 3, Dose Level 1 of Part 1b Combination Dose Escalation (SB 11285 combination with atezolizumab) will be opened for enrollment. After determination of MTD and RP2D in SB 11285 plus atezolizumab combination the Part 2 with Expansion Cohorts will commence to further evaluate the RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least ≥18 years of age (male or female).
2. Disease characteristics for patients in Part 1:

   a. Patient with any histologically or cytologically confirmed solid tumor that is locally advanced or metastatic or unresectable tumor and has disease progression after treatment with available therapies that are known to confer clinical benefit or who are intolerant to treatment.

   Note: Tumor types of primary interest in Part 1 Dose Escalation include tumors which are relapsed or refractory after anti PD-1/PD-L1 therapy (include but not limited to malignant melanoma, HNSCC, renal cell carcinoma, hepatocellular carcinoma, Merkel cell carcinoma, urothelial, non-small cell lung cancer, gastric carcinoma, ovarian carcinoma, endometrial, TNBC, cervical cancer, and colorectal carcinoma)
3. Disease characteristics and prior treatments for patients in Part 2:

   1. Cohort A (Melanoma): Patients with advanced or metastatic melanoma who have progressed following treatment with an anti-PD-1 or anti-PD-L1 antibody. Patients with BRAF mutated melanoma must have previously received BRAF/MEK targeted therapy.
   2. Cohort B (Head and Neck): Patient has anti-PD-1/PD-L1 refractory metastatic or recurrent HNSCC of the oral cavity, oropharynx, hypopharynx, or larynx. Participants may not have a primary tumor site of the nasopharynx (any histology).

   i. Has histologically confirmed Stage III, IVa, or IVb disease per TNM staging, American Joint Committee on Cancer (AJCC, 8th edition), with recurrent or persistent disease after definitive chemoradiation, deemed unresectable and considered refractory to both platinum-based combination chemotherapy and anti-PD-1/PD-L1 antibody therapy OR ii. Has histologically confirmed Stage IVc disease per TNM staging, AJCC 8th edition, considered refractory to platinum-based combination chemotherapy and anti-PD-1/PD-L1 antibody therapy.

   c. Cohort C: Tumor types not in Cohort A and B - Naïve or relapsed refractory to anti PD-1/PD-L1
4. An Eastern Cooperative Oncology Group (ECOG) performance status ≤1
5. Estimated life expectancy ≥3 months
6. Measurable disease according to RECIST criteria v 1.1
7. Patients must have recovered (ie, to NCI CTCAE grade ≤1) from all toxicity associated with previous treatments (exception: patients may enter with continuing alopecia irrespective of CTCAE grade).
8. All women of childbearing potential must have a negative pregnancy test at Screening, prior to study drug administration
9. Women of childbearing potential include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal. Postmenopausal is defined as: (1) Amenorrhea ≥12 consecutive months without another cause and a documented serum follicle stimulating hormone (FSH) level >35 mIU/mL; (2) Women with irregular menstrual periods and a documented serum FSH level >35 mIU/mL; or (3) Women on hormone replacement therapy (HRT)
10. All patients, male and female, who are not surgically sterilized or postmenopausal as defined above, must agree to use dual effective birth control during the study and for at least 28 days after the last dose of study medication and 5 months after the last dose of atezolizumab.

    Highly effective methods of contraception are hormonal contraceptives (oral, injectable, patch, intrauterine devices), male partner sterilization, or total abstinence from heterosexual intercourse, when this is the preferred and usual lifestyle of the patient. Note: The double-barrier method (eg, synthetic condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel), periodic abstinence (such as calendar, symptothermal, post-ovulation), withdrawal (coitus interruptus), lactational amenorrhea method, and spermicide only are not acceptable as highly effective methods of contraception
11. Patients has adequate hematologic and organ function, defined as:

    1. ANC ≥1500 mm3 without requiring G-CSF
    2. Platelets ≥100,000/mm3
    3. Hemoglobin ≥9 g/dL Note: Patients with Hb 7 to ≤9 g/dL (without bleeding) transfused prior to dosing in order to meet eligibility criteria
    4. Serum creatinine ≤1.5× upper limit of normal (ULN) for the reference laboratory or creatinine clearance ≥50 mL/min within the 28 days before enrollment (calculated from Cockcroft-Gault formula or 24 hour urine collection).
    5. Alanine aminotransferase (ALT), aspartate transaminase (AST) ≤3.0× the upper limit of normal (ULN) if no liver involvement or ≤5×ULN with liver involvement
    6. Adequate coagulation: prothrombin time (PT), an International Normalized Ratio (INR) or activated partial thromboplastin time (aPTT) ≤1.5×ULN or for patients requiring anticoagulant therapy, the PT/INR, aPTT should be within therapeutic range of the given anticoagulant agent
    7. Total bilirubin ≤1.5×ULN (or total serum bilirubin ≤3×ULN for patients with Gilbert's disease)
12. Patients must be willing and able to provide written informed consent prior to the performance of any study-specific procedure

Exclusion Criteria:

1. Women who are pregnant or lactating or expecting to conceive a child within the projected duration of the study
2. History or evidence of cardiovascular (CV) risk including any of the following: Recent (within the past 6 months) history of serious uncontrolled cardiac arrhythmia or clinically significant ECG abnormalities including second degree (Type II) or third degree atrioventricular block; Cardiomyopathy, myocardial infarction, acute coronary syndromes (including unstable angina pectoris), coronary angioplasty, stenting, or bypass grafting within the past 6 months before enrolment; Congestive heart failure (Class II, III, or IV) as defined by the New York Heart Association functional classification system (NYHA).
3. Patients with marked Baseline QTc prolongation (QT interval corrected for rate by Fridericia's formula [QTcF] ≥470 msec for women and ≥450 msec for men on the ECG obtained at Screening by mean of three ECGs).
4. Use of concomitant medications known to moderately or severly prolong QT interval.
5. Patients with active or ongoing infection requiring systemic IV antibiotic therapy. Patients with active or ongoing Epstein-Barr virus, hepatitis B virus, or hepatitis C virus or with known human immunodeficiency virus (HIV) infection, tuberculosis, or other infections within 4 weeks.
6. Clinically significant pulmonary disease, chronic or recurrent renal or urinary tract disease, liver disease, endocrine disorder, autoimmune disorder, or neuromuscular, musculoskeletal, or mucocutaneous conditions that, in the opinion of the Investigator, put the patient at additional risk by participating in the study or otherwise make the patient unsuitable for the study
7. The patient has uncontrolled intercurrent illness including, but not limited to uncontrolled infection, including uncontrolled diabetes mellitus or decreased pulmonary function, or psychiatric illness/social situations that would limit compliance with study
8. Has an active autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease modifying agents, corticosteroids, or immunosuppressive drugs) except vitiligo or resolved childhood asthma/atopy. Replacement therapy, such as thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, is not considered a form of systemic treatment
9. Patients with a history of or active pneumonitis Grade ≥ 2 (from any etiology).
10. Patients who have discontinued prior immunotherapy due to immune-related adverse reaction(s)
11. Is on chronic systemic steroid therapy in excess of replacement doses (prednisone ≤10 mg/day is acceptable), or on any other form of immunosuppressive medication. Note: The use of physiologic replacement doses of corticosteroids may be approved after consultation with the Sponsor's Medical Monitor or designee
12. Patients who have undergone major surgery within the last 4 weeks
13. Patients with new brain metastasis. Patients with treated (surgically excised or irradiated) and stable brain metastases are eligible as long as the treatment was at least 4 weeks prior to initiation of study drug and baseline brain CT with contrast or MRI within 2 weeks of initiation of study drug is negative for new brain metastases
14. Active malignant disease other than that being treated in this study. Exceptions: malignancies that were treated curatively and have not recurred within the past 2 years; completely resected basal cell carcinoma and squamous cell carcinoma of the skin; and completely resected carcinoma in situ of any type.
15. Patient- Prior treatment with the following agents:

    1. Stimulator of Interferon Genes (STING) agonist at any time.
    2. Anticancer therapy or investigational therapy within 28 days or 5 half-lives of the drug, whichever is shorter; "Check-point inhibitors", including Programmed death receptor-1 (PD-1), PD-L1 and Cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) inhibitors within 28 days (except part 2 Cohort C);
    3. Prior radiation therapy: permissible if at least 1 non-irradiated measurable lesion is available for assessment according to RECIST version 1.1 or if a solitary measurable lesion was irradiated, objective progression is documented. A wash out of at least 28 days before start of study treatment for radiation of any intended use to the extremities for bone metastases and 28 days for radiation to the chest, brain, or visceral organs is required. Palliative radiation is permissible at any time before or during the study.
16. Receipt of any live vaccines within 4 weeks prior to the initiation of study drug and anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab.
17. Patients considered by Investigators for any other reason to be unsuitable for the study or unable to comply with all study procedures and follow-up examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Part 1: Observation of DLT | Cycle 1 (4 weeks)
  Dose-limiting toxicity (DLT) is defined as a clinically significant adverse event or abnormal laboratory value occurring during Cycle 1 (Days 1-28) during both monotherapy and Combination dose-escalation portions of Part 1. Adverse events will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Part 1: Determination of the MTD | Cycle 1 (4 Weeks)
  The maximum tolerated dose (MTD) will be defined as the highest dose level below the maximum administered dose that has confirmed less than 2 out of 6 subjects with DLT. At least 6 subjects evaluable for the safety endpoint must be entered at this dose level before it may be confirmed as the MTD.
Part 1: Determination of the RP2D | 8 weeks to 12 months
  The recommended phase 2 dose (RP2D) will be based on a consideration of the totality of data including but not limited to safety data (including DLTs), PK, PD and preliminary efficacy, as available after completion of Part 1
Part 1: Incidence of Adverse Events [Safety and Tolerability] | 4 weeks to 12 months
  Incidence of adverse events of SB 11285 as a monotherapy and in combination with atezolizumab when administered as an IV infusion, as determined by patient reporting, clinical laboratory test changes from baseline (hematology, serum chemistry, coagulation, urinalysis, pregnancy, thyroid panel), and clinically significant changes in physical examination data (vital signs and ECG)
Part 2: Preliminary antitumor activity of SB 11285 in combination with atezolizumab | 28 Days to 12 months
  Preliminary antitumor activity of SB 11285 in combination with atezolizumab in patients with solid tumors, will be evaluated in terms of objective response rate as assessed by the Investigators using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and and by iRECIST
Part 2: Confirmation of recommended RP2D and schedule of SB 11285 in combination with atezolizumab | 4 weeks to 12 months
  Confirmation of the recommended phase 2 dosage (RP2D) and dosing interval will be based on consideration of the totality of available data, including safety, PK, PD, and preliminary efficacy, as available.
Part 2: Incidence of adverse events [Safety and Tolerability] | 4 Weeks to 12 months
  Incidence of adverse events of SB 11285 in combination with atezolizumab when administered as an IV infusion, as determined by patient reporting, clinical laboratory test changes from base line (hematology, serum chemistry, coagulation, urinalysis, pregnancy, thyroid panel), and clinically significant changes in physical examination data (vital signs and ECG)

SECONDARY OUTCOMES:
Part 1 and 2: Cmax (Plasma of SB 11285) | up to 12 months
  To characterize the plasma pharmacokinetics (PK) of SB 11285 following IV administration of SB 11285 as monotherapy and in combination with atezolizumab, the PK endpoint maximum plasma concentration (Cmax) will be measured.
Part 1 and 2: Time to Cmax (Plasma of SB 11285 ) | up to 12 months
  To characterize the plasma pharmacokinetics (PK) of SB 11285 following IV administration of SB 11285 as monotherapy and in combination with atezolizumab, the PK endpoints time to maximum plasma concentration (Cmax) will be measured.
Part 1 and 2: AUC (Plasma of SB 11285 ) | up to 12 months
  To characterize the plasma pharmacokinetics (PK) of SB 11285 following IV administration of SB 11285 as monotherapy and in combination with atezolizumab, the PK endpoint area under the concentration-time curve will be measured.
Part 1 and 2: Cmax (Plasma of SB 11312) | up to 12 months
  To characterize the plasma pharmacokinetics (PK) of SB 11312 following IV administration of SB 11285 as monotherapy and in combination with atezolizumab, the PK endpoint maximum plasma concentration (Cmax) will be measured.
Part 1 and 2: Time to Cmax (Plasma of SB 11312) | up to 12 months
  To characterize the plasma pharmacokinetics (PK) of SB 11312 following IV administration of SB 11285 as monotherapy and in combination with atezolizumab, the PK endpoints time to maximum plasma concentration (Cmax) will be measured.
Part 1 and 2: AUC (Plasma of SB 11312) | up to 12 months
  To characterize the plasma pharmacokinetics (PK) of SB 11312 following IV administration of SB 11285 as monotherapy and in combination with atezolizumab, the PK endpoint area under the concentration-time curve will be measured.
Part 1 and 2: Plasma of SB 11312 | up to 12 months
  To characterize the plasma pharmacokinetics (PK) of SB 11312 following IV administration of SB 11285 as monotherapy and in combination with atezolizumab, the PK endpoint area under the concentration-time curve will be measured.
Part 1: Objective response rate (ORR) | 4 weeks to 12 months
  Objective response rate (ORR) assessed by RECIST v 1.1 for patients in Part 1 only
Part 1 and 2: Duration of response (DOR) | 4 weeks to 12 months
  Duration of response (DOR) assessed by RECIST v 1.1 and by iRECIST (Part 1 and 2)
Part 1 and 2: Progression-free survival (PFS) | 4 weeks to 12 months
  Progression-free survival (PFS) assessed by RECIST v 1.1 and by iRECIST
Part 1 and 2: Overall survival (OS) | up to 39 months
  Overall survival (OS) is defined as time from date of first study treatment to death due to any cause. The Kaplan-Meier method will be used to estimate the median OS.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Laing, Study Director — Vice-President of Clinical Development
Locations (2):
- United States (2):
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania